CLINICAL TRIAL: NCT06946927
Title: A Phase Ib, Dose Escalation and Expansion Study to Evaluate the Safety, Tolerability, Pharmacokinetics and Efficacy of JMKX001899 in Combination With Other Therapies in Subjects With Locally Advanced or Metastatic Non-Small Cell Lung Cancer With KRAS G12C Mutation.
Brief Title: A Phase Ib Study of JMKX001899 in Combination With Other Therapies in Advanced NSCLC Harboring KRAS G12C Mutation
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jemincare (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: JMKX1899-C101
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-04

CONDITIONS: NSCLC (Advanced Non-small Cell Lung Cancer)
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung | interventions — Carboplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort A: JMKX001899+IN10018 (Experimental)
  Interventions: Drug: JMKX001899; Drug: IN10018
- Cohort B: JMKX001899+chemotherapy (Experimental)
  Interventions: Drug: JMKX001899; Drug: Chemotherapy: Pemetrexed; Drug: Carboplatin
- Cohort C: JMKX001899+IN10018+chemotherapy (Experimental)
  Interventions: Drug: JMKX001899; Drug: IN10018; Drug: Chemotherapy: Pemetrexed; Drug: Carboplatin

INTERVENTIONS:
Drug: JMKX001899 — JMKX001899 tablet administered orally daily.
Drug: IN10018 — IN10018 tablet administered orally daily.
  Arms: Cohort A: JMKX001899+IN10018; Cohort C: JMKX001899+IN10018+chemotherapy
Drug: Chemotherapy: Pemetrexed — IV infusion once every 3 weeks
  Arms: Cohort B: JMKX001899+chemotherapy; Cohort C: JMKX001899+IN10018+chemotherapy
Drug: Carboplatin — IV infusion once every 3 weeks, 4 Cycles
  Arms: Cohort B: JMKX001899+chemotherapy; Cohort C: JMKX001899+IN10018+chemotherapy

SUMMARY:
This is a phase 1b, dose escalation and expansion study to evaluate the safety, tolerability, pharmacokinetics and efficacy of JMKX001899 in combination with IN10018 or in combination with chemotherapy or in combination with IN10018 and chemotherapy in subjects with locally advanced or metastatic NSCLC with KRAS G12C mutation.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically documented Stage IIIB or IIIC NSCLC disease not amenable for surgical resection or definitive chemoradiation or Stage IV NSCLC disease.
2. Known KRAS G12C mutation, and negative results for other driver genes with approved targeted therapies.
3. Measurable disease according to RECIST 1.1.
4. An Eastern Cooperative Group (ECOG) performance status of 0 or 1.
5. Adequate organ function.

Exclusion Criteria:

1. Subjects with carcinomatous meningitis or spinal cord compression; or with other evidence indicating that central nervous system (CNS) metastases or leptomeningeal metastases are not yet controlled.
2. Prior chemotherapy, radiotherapy, immunotherapy or treatment with an investigational agent within 4 weeks of receipt of study drug (within 6 weeks for nitrosoureas, mitomycin C; within 2 weeks of small molecule targeted therapies, traditional medicine with anticancer indication).
3. History of prior malignancy in the past 3 years, with the exception of curatively treated malignancies.
4. Gastrointestinal (GI) tract disease causing the inability to take oral medication or affect drug absorption.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 72 (Estimated)
Dates: Start 2025-06-06 (Actual); Primary Completion 2026-02 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II dose (RP2D) | approximately 1 year
adverse events | Through study completion, approximately 2.5 years

CONTACTS AND LOCATIONS:
Overall Officials: Yilong Wu, Principal Investigator — Guangdong Provincial People's Hospital
Locations (1):
- Guangdong Provincial People's Hospital, Guangzhou, Guangdong, China